CLINICAL TRIAL: NCT02071186
Title: The Effect of Non-pharmacological Novel Cognitive Interventions on Motor-Cognitive Function in Children With Attention Deficit Hyperactivity Disorder
Brief Title: The Effect of Non-pharmacological Novel Cognitive Interventions on Motor-Cognitive Function in Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-13-YL-0544-CTIL
Record Dates: First submitted 2014-02-15; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Virtual Reality training (Experimental): Subjects will be asked to walk on a treadmill while negotiating virtual obstacles. The VR system includes a camera based motion capture and a computer generated simulation. The camera is used to capture the movement of the participant's feet. These images are then transferred to the computer simulation and projected to the patient on a screen. The speed, orientation, size, frequency of appearance and shape of the targets are manipulated to increase task difficulty. The Virtual environment imposes a cognitive load requiring attention and response selection as well as processing of rich visual stimuli involving several perceptual processes. The system provides visual and auditory feedback of task performance to enhance motor learning.
  Interventions: Device: Virtual Reality training
- Computerized Cognitive Remediation (Experimental): The "AttenGo" program will be used for neuro-cognitive remediation aimed at enhancing attention, concentration, working memory, and executive function. The program has shown to be effective in improving attention and executive function in children with ADHD. The training is composed of cognitive exercises that challenge subjects with problem solving, information processing, response inhibition and dividing attention. The users receive immediate feedback from the system when losing focus. The program is adaptive and progresses according to the subjects abilities.
  Interventions: Other: Computerized Cognitive Remediation
- Control group (Active Comparator): Subjects in this group will be assessed based on the study protocol but will receive no treatment other than their standard of care which could include pharmacological or/ and non-pharmacological treatment.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Virtual Reality training — Subjects will train with the VR system at the Tel Aviv Sourasky Medical Center 3 times per week for 6 weeks with each session lasting approximately 30 minutes.
  To assure participants' safety and maintaining progress, training with the VR will be individual and provided by qualified physiotherapists, who use the system on a daily basis.
  Arms: Virtual Reality training
Other: Computerized Cognitive Remediation — Subjects in this study will train with the AttenGo program at home 3-5 times per week for 6 weeks with each session lasting approximately 30 minutes.
  Arms: Computerized Cognitive Remediation
Other: Standard of care
  Arms: Control group

SUMMARY:
The purpose of this study is to test the hypothesis that cognitive remediation and virtual reality treatment approaches can enhance cognitive and motor function in children with ADHD.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is the most common neurobehavioral disorder affecting children. ADHD is currently treated with a combination of medication and behavioral therapy aimed at reducing the negative symptoms. Pharmacologic treatment methods, such as the use of Methylphenidate (MPH) have many drawbacks including high cost and side effects.

Non-pharmacological treatment approaches teach strategies aimed at improving behavior and environmental management. Evidence on efficacy of these treatments is lacking and the literature only supports the 'parental education' approach.

Motor aspects of the disorder tend to be undertreated. Studies have shown that persistent use of MPH has a positive effect on motor output timing and coordination in children with ADHD. Thus non-pharmacological interventions aimed at improving attention are likely to also improve other aspects of the disorder such as motor problems and thus should be further explored.

Various computerized remediation programs have been developed as a non-pharmacological alternative for children with ADHD. The programs present exercises that require sustained attention and a response to set rules and are often graded in task complexity according to the user's abilities.

Virtual Reality (VR) is a simulation of the real world using computer graphics that requires interaction, immersion and active participation by the user. VR applications have shown to be effective in improving attention in children and adolescents with behavioral problems, teaching them to focus on some tasks more than existing cognitive training programs. VR while walking has demonstrated improvements in both motor and cognitive function in older adults and patients with neurodegenerative diseases suggesting a beneficial effect on motor and cognitive function. However this treatment has not been tested yet in ADHD.

The study will investigate the following aims:

1. To compare the effect of computerized cognitive remediation and VR on attention and gait in children with ADHD.
2. To examine the long term effects of computerized cognitive remediation and VR on attention and gait in children with ADHD.
3. To compare, in an exploratory analysis, the effects of the non-pharmacological training paradigms to standard of care treatment on attention and gait in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with ADHD by a pediatrician, child neurologist or child psychiatrist, according to the ADHD criteria in the Diagnostic and Statistical Manual of Mental Disorders 5th edition.
* Attending regular education frameworks
* Have access to a personal computer at home

Exclusion Criteria:

* Children on active medication for ADHD during the study period
* Are taking any other medication that could affect attention, balance or motor function
* Have a serious medical condition that could affect attention, gait or balance
* Have any known genetic syndromes, autism, neurological conditions or psychiatric disorders or any medical illness requiring immediate treatment
* Are participating in a competing exercise program designed to improve gait or balance

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Immediate change in gait function | One week post intervention
  Gait speed and variability will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance.
Immediate change in cognitive function | One week post intervention
  A computerized neuropsychological test battery will be used to assess different cognitive domains including memory, attention, executive function, visual spatial processing and a global cognitive composite score. These measures will be compared to baseline performance.

SECONDARY OUTCOMES:
Retention of change in gait function | One month post intervention
  Gait speed and variability will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared performance at baseline and at one week post intervention.
Retention of change in cognitive function | One month post intervention
  A computerized neuropsychological test battery will be used to assess different cognitive domains including memory, attention, executive function, visual spatial processing and a global cognitive composite score. These measures will be compared performance at baseline and at one week post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Leitner, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel